CLINICAL TRIAL: NCT01351558
Title: Exercise and Alterations in Pain Sensitivity
Brief Title: Exercise and Pain Sensitivity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties.
Sponsor: Henning Bliddal (Other)
Responsible Party: Sponsor-Investigator, Henning Bliddal, Professor, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 101.01; 10-093704 (Other Grant/Funding Number: Danish Research Council)
Record Dates: First submitted 2011-05-09; First posted 2011-05-11 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Knee Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (No Intervention): No intervention for 12 weeks
- Knee muscle strengthening exercises (Active Comparator)
  Interventions: Other: Knee muscle strengthening exercises
- Upper extremity strengthening exercises (Active Comparator)
  Interventions: Other: Upper extremity strengthening exercises
- Cardiovascular fitness exercises (Active Comparator)
  Interventions: Other: Cardiovascular fitness exercises

INTERVENTIONS:
Other: Knee muscle strengthening exercises — Muscle strengthening exercises of the quadriceps and hamstring muscles will be performed based on a standard muscle strengthening exercise paradigm: 3 sets with 6-8 repetitions (corresponding to approximately 80% repetition maximum (RM)) will be performed. The training load will be progressed by means of weekly estimates of muscle strength to ensure a constant load of 80% RM. The exercises will be supervised
  Arms: Knee muscle strengthening exercises
Other: Upper extremity strengthening exercises — Muscle strengthening exercises of the upper amrs and shoulder girdle will be performed based on a standard muscle strengthening exercise paradigm: 3 sets with 6-8 repetitions (corresponding to approximately 80% repetition maximum (RM)) will be performed. The training load will be progressed by means of weekly estimates of muscle strength to ensure a constant load of 80% RM. The exercises will be supervised
  Arms: Upper extremity strengthening exercises
Other: Cardiovascular fitness exercises — Cardiovascular fitness exercises encompass circuit training including exercises on (but not limited to): ergometer cycles, treadmills (running), and cross-trainers. The exercise intensity is aiming at exercises within 60-85% of maximum heart rate (defined as 220 - age). The heart rate is monitored using a standard heart rate monitor. The exercises will be supervised
  Arms: Cardiovascular fitness exercises

SUMMARY:
There is ample evidence that exercise therapy is beneficial with respect to pain in patients with osteoarthritis of the knee. However, the pain relieving mechanisms are unknown. To enhance the efficacy of exercise therapy a deeper understanding of the involved mechanisms is needed.

Different exercise types may affect the pain sensitivity differently. It is hypothesized that non-specific exercises (i.e. exercises that does not involve the knee) reduces the processing of pain in the central nervous system (central sensitivity) to knee joint pain in healthy subjects. It is also hypothesized that exercises that involve the knee (i.e. specific knee exercises) reduce the sensitivity of pain receptors in the knee (peripheral sensitivity) in healthy subjects.

Healthy volunteers are recruited and randomised to one of four interventions: 1: Muscle strengthening exercises involving the thigh muscles; 2: Muscle strengthening exercises involving the shoulder muscles; 3: Cardio-vascular fitness exercises; or 4: Control (no exercises). The active interventions include exercises three times per week for 12 weeks. Pain sensitivity and a range of explanatory variables is measured before the interventions, after 4 weeks and after 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 35 years
* Untrained (i.e. less than 2 hours of organised exercise per week in the last 6 months - physical activity related to transportation (e.g. bicycling) is not included)
* Generally healthy according a medical exam at screening, history
* Willing and able to participate in all measurements
* Willing and able to attend all training sessions
* Willing to keep the habitual activity and amount of training constant (ie screening activity and training volume).
* 20 ≤ body mass index (BMI) ≤ 28 kg/m2
* Speak, read and write Danish

Exclusion Criteria:

* Pregnant or breastfeeding
* Current or previous symptoms of autoimmune disease (eg, inflammatory bowel disease, multiple sclerosis, lupus, rheumatoid arthritis)
* Planned surgery during the study period
* Current or former musculoskeletal injuries or illnesses, including but not confined to:
* Ligament Injuries
* Meniscus Injuries
* Osteoarthritis
* Patellofemoral Pain Syndrome
* Backache
* Neck pain
* tendinopathy
* Current or past diagnosis, signs or symptoms of significant cardiovascular disease, including but not limited to:
* Ischemic heart disease
* Arteriosclerosis
* Medical conditions that contraindicate exercise, including but not limited to:
* Chronic or congenital heart disease
* Asthma
* Chronic Obstructive Pulmonary Disease
* Past or current diagnosis, signs or symptoms of significant neurological disease, in-incl. but not limited to:
* Blood clot in brain
* Stroke
* Clinically significant head trauma within the last year
* Peripheral neuropathy
* Epilepsy or seizures
* Impaired balance
* Alcohol or drug abuse within the past 5 years
* Past or current diagnosis, signs or symptoms of major psychiatric disorder
* Regional pain syndromes like fibromyalgia
* Regional pain caused by lumbar nerve root or cervical radiculopathy with or at risk for developing it

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2011-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change in pressure pain sensitivity | Baseline, and after 12 weeks of exercise

SECONDARY OUTCOMES:
Change in muscle strength | baseline and after 12 weeks
  Muscle strength is measured in knee extension and flexion and in arm extension and flexion (bench press and pull)
Change in cardiovascular fitness | baseline after 4 weeks and after 12 weeks
  Watt max test is performed on a bicycle ergometer to estimate the maximal oxygen uptake velocity
Change in baroreflex sensitivity | baseline after 4 weeks and after 12 weeks
  Heart rate and blood pressure variability is measured during rest and during quiet standing.

CONTACTS AND LOCATIONS:
Overall Officials: Marius Henriksen, PT,PhD, Principal Investigator — Senior Researcher
Locations (1):
- The Parker Institute, Frederiksberg University Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Henriksen M, Klokker L, Bartholdy C, Graven-Nielsen T, Bliddal H. The Associations between Pain Sensitivity and Knee Muscle Strength in Healthy Volunteers: A Cross-Sectional Study. Pain Res Treat. 2013;2013:787054. doi: 10.1155/2013/787054. Epub 2013 Sep 17. PMID 24167727